CLINICAL TRIAL: NCT00076518
Title: A Phase II Trial of the Effect of Combination Therapy With Fish Oil Supplement and Fenofibrate on Triglyceride (TG) Levels in Subjects on Highly Active Antiretroviral Therapy (HAART) Who Are Not Responding to Either Fish Oil or Fenofibrate Alone
Brief Title: The Effect of Fish Oil Plus Fenofibrate on Triglyceride Levels in People Taking Highly Active Antiretroviral Therapy (HAART)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5186; 10686 (Registry Identifier: DAIDS ES); ACTG A5186
Record Dates: First submitted 2004-01-26; First posted 2004-02-04 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hypertriglyceridemia
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hypertriglyceridemia | interventions — Fenofibrate; Fish Oils

INTERVENTIONS:
Drug: Fenofibrate
Drug: Fish Oil

SUMMARY:
The purpose of this study is to determine the effectiveness of fish oil supplements combined with the drug fenofibrate in treating elevated triglyceride levels in people taking anti-HIV drugs. The participants in this study will have shown no response to fish oil supplements or fenofibrate alone.

DETAILED DESCRIPTION:
Although highly active antiretroviral therapy (HAART) has decreased the morbidity and mortality caused by HIV infection, its use has been associated with lipid abnormalities, particularly elevations in serum triglycerides. Hypertriglyceridemia is a risk factor in the development of cardiovascular and cerebrovascular disease as well as pancreatitis. Lipid-lowering drugs called fibrates have been part of the recommended treatment for elevated triglycerides, but the response to fibrates is incomplete in a large proportion of people. Fish oil capsules containing large amounts of omega-3 fatty acids have been shown to decrease serum triglycerides. However, fish oil supplements or fibrates alone are often inadequate for treating hypertriglyceridemia in people taking HAART. This study will determine whether the combination of the two therapies will lower serum triglycerides in people on HAART more effectively than either therapy alone.

This study comprises two steps. In Step I, participants will be randomly assigned to receive either fish oil supplements or fenofibrate. Participants will be evaluated for treatment response at Week 8. Those who have responded to their treatment will remain on their original single agent therapy through Week 18. Those who have not responded to treatment at Week 10 will move on to Step 2 and begin combination therapy with both fenofibrate and fish oil until Week 18. All participants will return at Week 22 for a follow-up visit. Except at the Week 10 visit, participants will be expected to fast prior to all study visits. Participants will remain on their individual HAART regimens for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Fasting LDL <= 160 mg/dL and fasting serum triglycerides >= 400 mg/dL within 28 days prior to study entry
* Willing and able to adhere to a lipid-lowering diet and exercise program for at least 28 days prior to study start and for the duration of the study
* Treatment with HAART for at least 3 months prior to study entry. Participants must be on stable HAART for at least 4 weeks immediately prior to study entry. Participants who have changed from a protease inhibitor (PI)-based regimen to a non-PI-based regimen in the previous 3 months must be on stable HAART for at least 8 weeks immediately prior to study entry.
* Willingness to remain on current HAART regimen for the duration of the study
* Women of reproductive potential must use an acceptable method of contraception while receiving study drugs and for at least 4 weeks after stopping the study drugs
* Men on testosterone replacement therapy must have been on stable therapy for at least 3 months prior to study entry and must be willing to continue stable therapy for the duration of the study
* Participants on hormone replacement therapy other than testosterone replacement therapy and participants using oral contraceptives must have been on stable therapy for at least 28 days prior to study entry and must be willing to continue stable therapy for the duration of the study

Exclusion Criteria:

* Use of investigational antiretroviral drugs within 28 days prior to study entry. Investigational therapies allowed by the study chairs or given in an AACTG study or expanded access trial are permitted, as long as the treatment can be continued for the duration of this study.
* Coronary heart disease
* Atherosclerotic disease risk
* Congestive heart failure
* Uncontrolled hypertension within 28 days prior to study entry
* Active bleeding disorder or active peptic ulcer disease
* Diabetes mellitus that requires pharmacological, dietary control, or diabetic medication within 28 days prior to study entry
* Untreated hypothyroidism. Participants who are currently being treated for hypothyroidism are not excluded if the treatment was initiated at least 28 days prior to study entry.
* Use of levothyroxine or liothyronine, except for treatment of hypothyroidism, within 90 days prior to study entry.
* Active or symptomatic gallbladder disease within 1 year prior to study entry
* Use of systemic cancer chemotherapy within 60 days prior to study entry
* Cancer within 5 years prior to study entry. Skin cancers not requiring systemic treatment are allowed.
* Pregnancy or breast-feeding
* Use of any lipid-lowering agent within 28 days prior to study entry
* Use of hormonal anabolic therapies within 6 months prior to study entry
* Use of systemic steroids
* Use of immune modulators within 28 days prior to study entry
* Use of anticoagulants within 14 days prior to study entry
* Allergy or sensitivity to study drugs or their formulations
* Active drug or alcohol use or dependence that would interfere with adherence to study requirements
* Decreased mental capacity that would interfere with adherence to study requirements
* Active AIDS-defining opportunistic infection (OI) within 28 days prior to study entry. Participants who have no evidence of active disease and are receiving maintenance therapy for AIDS-related OIs will be eligible.
* Any acute illness within 28 days prior to study entry that would interfere with participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John G. Gerber, MD, Study Chair — University of Colorado Health Science Center
Locations (5):
- United States (5):
  - Ucsf Aids Crs, San Francisco, California
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island

REFERENCES:
- [Background] Mulligan K, Grunfeld C, Tai VW, Algren H, Pang M, Chernoff DN, Lo JC, Schambelan M. Hyperlipidemia and insulin resistance are induced by protease inhibitors independent of changes in body composition in patients with HIV infection. J Acquir Immune Defic Syndr. 2000 Jan 1;23(1):35-43. doi: 10.1097/00126334-200001010-00005. PMID 10708054
- [Background] Bonnet F, Bonarek M, De Witte S, Beylot J, Morlat P. Efavirenz-associated severe hyperlipidemia. Clin Infect Dis. 2002 Sep 15;35(6):776-7. doi: 10.1086/342326. No abstract available. PMID 12203183
- [Background] Phillipson BE, Rothrock DW, Connor WE, Harris WS, Illingworth DR. Reduction of plasma lipids, lipoproteins, and apoproteins by dietary fish oils in patients with hypertriglyceridemia. N Engl J Med. 1985 May 9;312(19):1210-6. doi: 10.1056/NEJM198505093121902. PMID 3990714
- [Background] Harris WS. Nonpharmacologic treatment of hypertriglyceridemia: focus on fish oils. Clin Cardiol. 1999 Jun;22(6 Suppl):II40-3. doi: 10.1002/clc.4960221408. PMID 10376196
- [Background] Pichard C, Sudre P, Karsegard V, Yerly S, Slosman DO, Delley V, Perrin L, Hirschel B. A randomized double-blind controlled study of 6 months of oral nutritional supplementation with arginine and omega-3 fatty acids in HIV-infected patients. Swiss HIV Cohort Study. AIDS. 1998 Jan 1;12(1):53-63. doi: 10.1097/00002030-199801000-00007. PMID 9456255
- [Derived] Gerber JG, Kitch DW, Fichtenbaum CJ, Zackin RA, Charles S, Hogg E, Acosta EP, Connick E, Wohl D, Kojic EM, Benson CA, Aberg JA. Fish oil and fenofibrate for the treatment of hypertriglyceridemia in HIV-infected subjects on antiretroviral therapy: results of ACTG A5186. J Acquir Immune Defic Syndr. 2008 Apr 1;47(4):459-66. doi: 10.1097/QAI.0b013e31815bace2. PMID 17971707